CLINICAL TRIAL: NCT07103525
Title: INSPIRE: Initiative for Chinese Sex Workers to Promote Wellbeing and Improve HIV Prevention by Reducing intersEctional Stigma
Brief Title: Initiative for Chinese Sex Workers to Promote Wellbeing and Improve HIV Prevention by Reducing intersEctional Stigma
Acronym: INSPIRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-01572; R34MH136914-01A1 (NIH)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: HIV Prevention; Wellbeing
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Female Sex Workers (FSWs) randomized to receive the intervention.
  Interventions: Behavioral: INSPIRE Initiative
- Control Group (Active Comparator): Female Sex Workers (FSWs) randomized to the control group.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: INSPIRE Initiative — Culturally relevant, multi-level intervention designed to increase HIV testing through reducing intersectional stigma. Intervention includes series of four one-on-one conversations (45 minutes each over a six-week period) via mobile phone between the Hunter peer advocates and FSWs, which are reinforced through weekly text messages from the peer advocates and through role-model stories shared online.
  Arms: Intervention Group
Behavioral: Standard of Care — Standard HIV prevention information with no tailored components via one mobile phone verbal conversation with peer advocates.
  Arms: Control Group

SUMMARY:
During the development phase (Aim 1), investigators will use a community-driven process to further refine a preliminary intervention design that was developed based on previous research.

For the intervention phase (Aim 2), investigators will conduct a pilot randomized controlled trial of the multi-level intervention. For the individual-level component of the intervention, investigators will recruit 70 Chinese immigrant FSWs who work in MPs in Queens, NYC (n=35 intervention participants and n=35 control participants).

To assess the feasibility and acceptability of intervention implementation (Aim 3), investigators will conduct in-depth qualitative interviews with 12 FSW study participants and the 2 peer advocates and focus groups with 4-5 staff from each of the 3 organizations (3 focus groups total and 12-15 focus group participants in total).

ELIGIBILITY:
Inclusion Criteria:

* Female Sex Workers: A person who identifies as a woman, Chinese, a massage parlor (MP) worker in Queens, who is at least 18 years old, and has provided sexual services in the past 12 months, will be eligible.
* Community advisory board (CAB) members: self identifies as a community member providing services to immigrant Chinese women and is at least 18 years old.
* Peer Advocates: self identifies as current or previous sex worker, is a Chinese adult woman, and speaks both Mandarin and English.
* Medical Providers: self identifies as a current medical provider who works with Chinese immigrant adults and speaks English.

Exclusion Criteria:

* Female Sex Workers: Because completion of HIV testing is our primary study outcome, women who received an HIV test in the previous 3 months or who know they are HIV-positive will be excluded from the study.
* Community advisory board (CAB) members: Does not speak English or is under the age of 18.
* Peer Advocates: Does not speak English/Mandarin or is under the age of 18.
* Medical Providers: Does not speak English or does not provide care to Chinese immigrant adults (e.g., pediatricians).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Completed HIV Testing | Follow-Up Visit 1 (Approximately Week 6)
  Assessed via self-report.

SECONDARY OUTCOMES:
Percentage of Participants with PrEP Uptake | Follow-Up Visit 1 (Approximately Week 6)
  Assessed via self-report; percentage of participants who begin PrEP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sahnah Lim, PhD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - CUNY-Hunter College, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, will be shared. The study protocol, statistical analysis plan, informed consent form, clinical study report and analytic code will be shared. All data will be deposited to the NIMH Data Archive (NDA) starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates. Anyone who wishes to access the data for any purpose will be granted access. The research community will have access to data when the award ends. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. Investigators will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be deposited to the NIMH Data Archive (NDA) starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: The research community will have access to data when the award ends. As required by NDA, studies will also be created that contain the data used for every publication. Those studies will be shared when the pre-print is available. NDA studies have digital object identifiers (DOI) to aid in findability. We will include that DOI in relevant publications. NDA will make decisions about how long to preserve the data, but that data archive has not deleted any deposited data up to now.